CLINICAL TRIAL: NCT01617538
Title: Application of Contrast Enhance Ultrasound to Evaluate Hemodynamics Change in MCA With Moderate to Severe Stenosis After 24-week Atorvastatin Treatment
Brief Title: Application of Contrast Enhance Ultrasound to Evaluate Hemodynamics Change in MCA With Moderate to Severe Stenosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Xu, MD, Xu Bin, Capital Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WS1788891-22-CT25
Record Dates: First submitted 2012-06-04; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Stenosis
Keywords: atherosclerosis; stenosis; statin therapy; Signs and Symptoms; Circulatory; Change
MeSH Terms: conditions — Constriction, Pathologic; Atherosclerosis; Signs and Symptoms | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin (Experimental): 30 patients who had MCA infarction within 6 months prior to screening, and has not received any statins treatment before stroke.in this study ,we will give them atorvastatin 40mg treatment for 24 weeks and monitor and evaluate the change of intracranial hemodynamics after treatment.
  Interventions: Drug: atorvastatin
- compare (No Intervention): 30 patients who had MCA infarction within 6 months prior to screening, and has not received any statins treatment.we will monitor and evaluate the intracranial hemodynamics as a baseline.

INTERVENTIONS:
Drug: atorvastatin — 40mg per day,duration for 24 weeks
  Other Names: brand names :FIZER
  Arms: Atorvastatin

SUMMARY:
Objective:

To monitor and evaluate the change of intracranial hemodynamics and MCA stenosis after 24-week atorvastatin treatment using CEUS, CTA and DSA.

Study design:

Total 30 patients (60 arteries) will be enrolled in this study, who had MCA infarction within 6 months prior to screening, and has not received any statins treatment before stroke.

Eligible patient will receive atorvastatin 40mg treatment for 24 weeks. Hemodynamics changes and MCA stenosis will be evaluated using CEUS at baseline, 3-month,and 6-month. MCA stenosis, bloodstream velocity, as well as clinical symptoms will be assessed at each visit and compared to baseline.

DETAILED DESCRIPTION:
The cerebral infarction resulted from medially and heavily narrow MCA is determined by the three-type screen method .For the first screen cerebral infarction patients of MCA area who has the stroke or TIA history In 6 months are determined by the clinic stroke measure table,transstadial Doppler ultrasonography (TCD) carotid ultrasonography and skull CT. For the second the MAC area infarction and vessel narrow are determined by the skull magnetic resonance (MRI) and magnetic resonance vessel imaging (MRA) and the MCA trend bloodstream dynamics feature and narrow extent Are observed by the strengthened ultrasonography (CEVS) For the third, The MCA narrow extent is measured by the DSA test which is currently regarded as a gold standard and /or by the CTA .The atorvastatin 20mg Treatment is given to the patients who all use the antiplatelet medicine The clinic symptom improvement MCA narrow extent and bloodstream velocity are dynamically observed visited and analysed respectively at the basic line 3 and 6 months after treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients who had MCA infarction of unilateral with moderate to severe stenosis within 6 months prior to screening, and has not received any statins treatment before stroke.

Exclusion Criteria:

* With side of extracranial carotid artery 70-100% severe narrow or block
* Vertebrobasilar artery lesions caused by cerebral infarction
* Have rheumatic heart disease, the atrial fibrillation of heart disease, those who Cerebral hemorrhage patients
* Serious liver and kidney function is not complete patients.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Hemodynamics changes and MCA stenosis | given atorvastatin 40mg treatment for 24 weeks
  Hemodynamics changes will be evaluaed using CEUS at baseline, 3-month,and 6-month.in order to evaluate the effect of atorvastatin, we will compare the baseline with 3-month,and compare the baseline with 6-month.a statistic analysis of measure data is conducted by the group T test,which conducted by SAS 9.13 English edition .

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Qin, master, Study Director — science study Dept
Locations (1):
- FuXing Hospital,Capital Medicial University, Beijing, China